CLINICAL TRIAL: NCT05124808
Title: Intensive Glycemic Targets in Overweight and Obese Women With Gestational Diabetes Mellitus: A Multicenter Randomized Trial
Brief Title: Intensive Glycemic Targets in Overweight and Obese Women With Gestational Diabetes
Acronym: iGDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Pittsburgh (Other); University of Alabama at Birmingham (Other); University of Oklahoma (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Christina Scifres, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11435; R01HD101476 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-11-18 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes; Pregnancy, High Risk; Overweight and Obesity
MeSH Terms: conditions — Diabetes, Gestational; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive glycemic targets (Experimental): Participants in this arm will target a fasting blood glucose of <90 mg/dL and 1 hour post-prandial blood glucose values <120 mg/dL.
  Interventions: Other: Intensive glycemic targets
- Standard glycemic targets (Active Comparator): Participants in this arm will target a fasting blood glucose of <95 mg/dL and 1 hour post-prandial blood glucose values <140 mg/dL.
  Interventions: Other: Standard glycemic targets

INTERVENTIONS:
Other: Intensive glycemic targets — Fasting blood glucose <90 mg/dL, 1 hour post-prandial blood glucose <120 mg/dL
  Arms: Intensive glycemic targets
Other: Standard glycemic targets — Fasting blood glucose <95 mg/dL, 1 hour post-prandial blood glucose <140 mg/dL
  Arms: Standard glycemic targets

SUMMARY:
This is a multicenter randomized clinical trial of 828 overweight and obese individuals with gestational diabetes designed to compare standard to intensive glycemic targets.

DETAILED DESCRIPTION:
The prevalence of both obesity and gestational diabetes mellitus (GDM) have increased, and each is associated with adverse perinatal outcomes including fetal overgrowth, neonatal morbidity, hypertensive disorders of pregnancy, and cesarean delivery. Women with GDM who are also overweight and obese have higher rates of pregnancy complications when compared to normal weight women with GDM, which may occur in part due to suboptimal glycemic control. The current recommendations for glycemic targets in pregnant women with diabetes are not rigorously defined, and they far exceed the mean fasting (70.9 ±7.8 mg/dL) and 1 hour post- prandial (108.9 ± 12.9 mg/dL) glucose values in pregnant women without GDM. Our prior work demonstrated that use of intensive (fasting <90, 1 hr post-prandial <120 mg/dL) compared to standard (fasting <95 mg/dL, 1 hr post-prandial <140 mg/dL) glycemic targets resulted in improved glycemic control without increasing the risk for hypoglycemia. The Intensive Glycemic Targets in Overweight and Obese Women with Gestational Diabetes Mellitus: A Multicenter Randomized Trial (iGDM Trial) is a large, pragmatic randomized clinical trial designed to investigate the impact of intensive versus standard glycemic targets on perinatal outcomes in women with GDM who are overweight and obese. During the 5-year project period, a multidisciplinary team of investigators from 4 medical centers representing regions of the U.S. with high rates of obesity will randomize 828 overweight and obese women with GDM to either intensive or standard glycemic targets. The specific aims of this project are: 1) Determine the effectiveness of intensive glycemic targets in reducing the risk for neonatal composite morbidity and large for gestational age birthweight in overweight and obese women with GDM, 2) Assess the safety of intensive glycemic targets as measured by the frequency of maternal hypoglycemia in overweight and obese women with GDM, and 3) Evaluate the cost-effectiveness of intensive glycemic control compared with standard glycemic control as measured by the incremental cost per case of neonatal morbidity and LGA birth weight prevented and per Quality-adjusted Life-year. The expected outcome of this study is high-quality evidence on the effectiveness, safety, and cost-effectiveness of intensive glycemic targets in reducing adverse perinatal outcomes among overweight and obese women with GDM. If proven effective, use of intensive glycemic targets in overweight and obese women with GDM will have an important positive impact on the health of these high risk women and their infants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-45
* Singleton gestation
* Gestational age between 12 0/7-32 6/7 weeks' gestation with gestational diabetes diagnosed during this time frame using either a 50g 1-hr GCT ≥200 mg/dL or two or more abnormal values on a 100g OGTT using the Carpenter-Coustan Criteria
* Overweight or obese BMI at the first prenatal visit (BMI ≥25 kg/m2 or ≥23 kg/m2 in Asian Americans)

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Inability to communicate with members of the study team, despite the presence of an interpreter
* Planned delivery at a non-study affiliated hospital
* Known renal disease with a baseline creatinine >1.5 mg/dL
* Significant fetal anomalies diagnosed prior to study enrollment (these will include anomalies such as gastroschisis, spina bifida, complex congenital heart disease, or serious karyotypic anomalies that may lead to early delivery or increased risk of neonatal death)
* Oral or IV/IM steroid use within 7 days of study enrollment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 828 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with composite neonatal morbidity | Within 7 days of delivery
  Composite of large for gestational age birth weight, neonatal hypoglycemia, neonatal jaundice, and neonatal respiratory distress syndrome

SECONDARY OUTCOMES:
Number of participants with large for gestational age birth weight | Birth
  ≥90th percentile birth weight for gestational age, based on US birth weight normograms
Number of participants with neonatal hypoglycemia | Within 24 hours of delivery
  Blood glucose <40 mg/dL in the 1st 24 hours of life
Number of participants with neonatal jaundice | Within 7 days of delivery
  Documentation of need for phototherapy
Number of participants with respiratory distress syndrome | Within 7 days of delivery
  Signs of respiratory distress (tachypnea, grunting, nasal flaring, cyanosis) with an oxygen requirement within the first 24 hours of life and the presence of radiologic chest findings of hypoaeration and reticulogranular infiltrates or those needing immediate intubation for respiratory distress syndrome
Maternal hyperglycemia | From randomization to delivery
  Percent of maternal glucose values ≥120 and ≥140 mg/dL from randomization through delivery
Early maternal glycemic levels | 7 days after randomization
  Mean fasting and post-prandial values in the 7 days after randomization
Pre-delivery maternal glycemic levels | 14 days prior to delivery
  Mean fasting and post-prandial values in the 14 days prior to delivery
Glycemic levels during study enrollment | Up to 29 weeks
  Mean fasting and post-prandial glucose values from study enrollment until delivery
Episodes of maternal hypoglycemia | From randomization to delivery
  Percent of all glucose values <60 mg/dL
Number of episodes of symptomatic maternal hypoglycemia | From randomization to delivery
  Number of episodes of symptomatic hypoglycemia, episodes of symptomatic hypoglycemia requiring assistance
Number of participants with hypertensive disorders of pregnancy (gestational hypertension and pre-eclampsia) | From randomization up to 30 days after delivery
  Gestational hypertension
  • Requires systolic blood pressure ≥140 or diastolic blood pressure ≥90 mm Hg on two occasions at least for hours apart after 20 weeks of gestational in a woman with a previously normal blood pressure
  Pre-eclampsia
  * Requires systolic blood pressure ≥140 or diastolic blood pressure ≥90 mm Hg on two occasions at least for hours apart after 20 weeks of gestational in a women with a previously normal blood pressure and at least one of the following:69
  * Proteinuria (≥300 mg/24 hour timed collection, protein/creatinine ratio >0.3, or 2+ proteinuria on dipstick)
  * Thrombocytopenia (platelets<100,000)
  * Elevated blood concentrations of liver transaminases to twice normal concentration
  * Creatinine >1.1 mg/dL or a doubling of the serum creatinine concentration
  * Headache, blurry vision, or epigastric/RUQ pain
  * Pulmonary edema
  OR Systolic blood pressure of 160 mm Hg or diastolic blood pressure of 110 mg Hg or more
Number of participants with small for gestational age birth weight | Birth
  ≤10th percentile birth weight for gestational age, based on US birth weight normograms
Number of participants with cesarean delivery | Delivery
  Cesarean delivery for any indication
Number of participants with preterm birth <37 weeks | Delivery
  Gestational age at delivery <37 0/7 weeks (spontaneous or indicated)
Number of participants with shoulder dystocia | Delivery
  Documentation in the medical record of failure to deliver the fetal shoulder with gentle downward traction on the fetal head, requiring additional obstetric maneuvers to effect delivery, as documented by the delivery physician
Number of participants with NICU admission | Within 7 days of delivery
  Admission to the neonatal intensive care unit for any indication in the first 7 days of life
Infant adiposity | Within 72 hours of delivery
  Calculated using a flank skinfold

CONTACTS AND LOCATIONS:
Overall Officials: Christina Scifres, MD, Principal Investigator — Indiana University
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Indiana University, Indianapolis, Indiana
  - University of Oklahoma, Norman, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed and the investigators have published the main manuscripts regarding the outcomes of the trial, de-identified data will be made available by request. All requests will require review and approval by the investigators and the institutional regulatory committees.
Supporting Information: Study Protocol
Time Frame: Data will be available one year after study completion.
Access Criteria: Data access will be possible after approval of the request for data by the primary study team and after appropriate regulatory documents are in place.

REFERENCES:
- [Derived] Scifres CM, Battarbee AN, Feghali MN, Pierce S, Edwards RK, Smith EM, Guise D, Bhamidipalli S, Daggy J, Tuuli MG. Intensive glycaemic targets in overweight and obese individuals with gestational diabetes mellitus: clinical trial protocol for the iGDM study. BMJ Open. 2024 Feb 29;14(2):e082126. doi: 10.1136/bmjopen-2023-082126. PMID 38423770